CLINICAL TRIAL: NCT05003388
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Multiple Sclerosis
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for MS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-8-ATG-9-03
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; stem cell treatment
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of multiple sclerosis

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) can be a devastating disease. There is evidence that mesenchymal stem cell treatment is safe and efficacious for the treatment of MS. Patients with MS will receive a single intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells. The dose for the infusion will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease requiring chemotherapeutic drugs such as methotrexate, an autologous T Cell vaccine will be utilized created from the patient's own T cells obtained by apheresis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-06-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: Kurtzke Expanded Disability Status Scale (EDSS) | Four year follow-up
  EDSS is a scale to evaluate the function of the central nervous system. It will be completed for each follow up point

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Athens Beverly Hills Medical Group, Glyfada, Athens, Greece

REFERENCES:
- [Background] Meyer-Moock S, Feng YS, Maeurer M, Dippel FW, Kohlmann T. Systematic literature review and validity evaluation of the Expanded Disability Status Scale (EDSS) and the Multiple Sclerosis Functional Composite (MSFC) in patients with multiple sclerosis. BMC Neurol. 2014 Mar 25;14:58. doi: 10.1186/1471-2377-14-58. PMID 24666846
- [Background] Petrou P, Kassis I, Levin N, Paul F, Backner Y, Benoliel T, Oertel FC, Scheel M, Hallimi M, Yaghmour N, Hur TB, Ginzberg A, Levy Y, Abramsky O, Karussis D. Beneficial effects of autologous mesenchymal stem cell transplantation in active progressive multiple sclerosis. Brain. 2020 Dec 1;143(12):3574-3588. doi: 10.1093/brain/awaa333. PMID 33253391
- [Background] Riordan NH, Morales I, Fernandez G, Allen N, Fearnot NE, Leckrone ME, Markovich DJ, Mansfield D, Avila D, Patel AN, Kesari S, Paz Rodriguez J. Clinical feasibility of umbilical cord tissue-derived mesenchymal stem cells in the treatment of multiple sclerosis. J Transl Med. 2018 Mar 9;16(1):57. doi: 10.1186/s12967-018-1433-7. PMID 29523171
- [Background] Li JF, Zhang DJ, Geng T, Chen L, Huang H, Yin HL, Zhang YZ, Lou JY, Cao B, Wang YL. The potential of human umbilical cord-derived mesenchymal stem cells as a novel cellular therapy for multiple sclerosis. Cell Transplant. 2014;23 Suppl 1:S113-22. doi: 10.3727/096368914X685005. Epub 2014 Nov 5. PMID 25385295